CLINICAL TRIAL: NCT00122343
Title: A Phase II Study of AP23573, an mTOR Inhibitor, in Female Adult Patients With Recurrent or Persistent Endometrial Cancer
Brief Title: AP23573 in Female Adult Patients With Recurrent or Persistent Endometrial Cancer (8669-019)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-019; AP23573-04-203
Record Dates: First submitted 2005-07-21; First posted 2005-07-22 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Endometrial Cancer
Keywords: Endometrial; Cancer
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms | interventions — ridaforolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): AP23573 will be administered intravenously (IV) at a fixed dose of 12.5 mg over 30 minutes once daily for 5 days (QDx5) every 2 weeks. A 4-week period comprised of 2 courses of AP23573 is defined as a cycle of treatment.
  Interventions: Drug: ridaforolimus

INTERVENTIONS:
Drug: ridaforolimus — AP23573 will be administered intravenously (IV) at a fixed dose of 12.5 mg over 30 minutes once daily for 5 days (QDx5) every 2 weeks. A 4-week period comprised of 2 courses of AP23573 is defined as a cycle of treatment.
  Other Names: deforolimus; AP23573; MK-8669; ridaforolimus was also known as deforolimus until May 2009

SUMMARY:
This is an open-label nonrandomized multi-center study designed to evaluate the effect of AP23573 in patients with recurrent or persistent endometrial cancer. The primary objective is to assess the efficacy of AP23573 in patients with recurrent or persistent endometrial cancer when administered once daily for 5 consecutive days (QDx5) every two weeks at a dose of 12.5 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age with histologically confirmed endometrial cancer
* Documented progression of endometrial cancer (e.g., within the last 3 months)
* If of childbearing potential, must agree to use approved barrier methods of contraception (non hormonal methods)
* Presence of at least one measurable lesion that can be accurately measured in at least one dimension with longest diameter ≥20 mm using conventional techniques or ≥10 mm with spiral computed tomography (CT) scan (or otherwise at least twice the reconstruction interval for CT or magnetic resonance imaging [MRI] scans). Previously irradiated lesions may be considered to be measurable provided: *there has been documented progression of the lesion(s) since completion of radiotherapy; and *the criteria for measurability as outlined above are met.
* ECOG performance status ≤ 2
* Minimum life expectancy of 3 months
* Adequate renal and hepatic function, defined as:

  * Total serum bilirubin ≤ 1.5 x ULN for the institution;
  * AST and/or ALT ≤ 2 x ULN for the institution;
  * Alkaline phosphatase < 1.5 x ULN for the institution (if > 1.5 x ULN, then alkaline phosphatase liver fraction must be < 1.5 ULN);
  * Serum albumin ≥ 2.5 g/dL;
  * Serum creatinine ≤ 1.5 x ULN for the institution.
* Adequate bone marrow function, defined as:

  * ANC ≥ 1.5 x 10^9/L;
  * Platelet count ≥ 100 x 10^9/L.
* Serum cholesterol <350 mg/dL and triglycerides < 400 mg/dL
* Able to understand and give written informed consent

Exclusion Criteria:

* Women who are pregnant or lactating
* Presence of brain metastases
* More than 2 prior regimens of cytotoxic chemotherapy or enzyme inhibitor therapy
* Prior therapy with rapamycin, rapamycin analogues or tacrolimus; or known sensitivity to these agents
* Anticancer treatment (chemotherapy, radiotherapy, immunotherapy, biological response modifiers, signal transduction inhibitors, etc.) within 4 weeks prior to the first dose of AP23573. The interval may be ≥ 2 weeks for hormonal therapy or signal transduction inhibitors with a half-life known to be <24 hours and must be ≥ 6 weeks for nitrosourea or mitomycin.
* Ongoing toxicity associated with prior anticancer therapy (except peripheral neuropathy of ≤ Grade 1 by National Cancer Institute [NCI] toxicity criteria)
* Another primary malignancy within the past three years (except for non-melanoma skin cancer and cervical carcinoma in situ)
* Known or suspected hypersensitivity to drugs formulated with polysorbate 80 (Tween) or any other excipient contained in the study drug
* Known Grade 3 or 4 hypersensitivity to macrolide antibiotics (e.g., clarithromycin, erythromycin, azithromycin)
* Significant uncontrolled cardiovascular disease
* Active infection requiring systemic therapy
* Known HIV infection
* Treatment with any investigational agent within 4 weeks prior to the first dose of AP23573
* Concurrent treatment with immunosuppressive agents other than prescribed corticosteroids at stable doses for ≥ 2 weeks prior to first planned dose of study drug. Nasal, ophthalmic, and topical glucocorticoid preparations are allowed as well as low dose maintenance steroid therapy for other conditions. Physiologic hormone replacement therapy (e.g., thyroid supplementation for thyroid deficiency or oral replacement glucocorticoid therapy for adrenal insufficiency) is allowed.
* Inadequate recovery from any prior surgical procedure or having undergone any major surgical procedure within 2 weeks prior to the first dose of AP23573. Patients who have recovered from placement of a central venous access port within 2 weeks of Cycle 1, Day 1 will be considered eligible.
* Presence of any other life-threatening illness or organ system dysfunction which, in the opinion of the Investigator, would either compromise the patient's safety or interfere with evaluating the safety of the study drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to assess the efficacy of AP23573 in patients with recurrent or persistent endometrial cancer when administered once daily for 5 consecutive days (QDx5) every two weeks at a dose of 12.5 mg/day. | Duration of the study

SECONDARY OUTCOMES:
Assess the safety and tolerability of this study drug regimen in this patient population | Duration of the study
Evaluate secondary efficacy endpoints of time to tumor progression, progression-free survival and duration of response | Duration of the study
Examine pharmacokinetic characteristics of AP23573 | Duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Frank Haluska, M.D., Ph.D., Study Chair — Ariad Pharmaceuticals

REFERENCES:
- [Result] Colombo N, McMeekin DS, Schwartz PE, Sessa C, Gehrig PA, Holloway R, Braly P, Matei D, Morosky A, Dodion PF, Einstein MH, Haluska F. Ridaforolimus as a single agent in advanced endometrial cancer: results of a single-arm, phase 2 trial. Br J Cancer. 2013 Mar 19;108(5):1021-6. doi: 10.1038/bjc.2013.59. Epub 2013 Feb 12. PMID 23403817